CLINICAL TRIAL: NCT01754519
Title: Phase II Trial of Single Fraction Radiation Therapy (SFRT) at Roswell Park Cancer Institute for Select Patients With Early Stage Breast Cancer
Brief Title: Radiation Therapy in Treating Post-Menopausal Women With Early Stage Breast Cancer Undergoing Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IDE not submitted
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cianna Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 108907; NCI-2009-01568 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 108907 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2012-11-23; First posted 2012-12-21 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Ductal Breast Carcinoma In Situ; Estrogen Receptor Negative; Estrogen Receptor Positive; HER2/Neu Negative; Invasive Cribriform Breast Carcinoma; Invasive Ductal Carcinoma, Not Otherwise Specified; Lobular Breast Carcinoma In Situ; Mucinous Breast Carcinoma; Papillary Breast Carcinoma; Progesterone Receptor Positive; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIC Breast Cancer; Tubular Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (radiation therapy) (Experimental): Patients undergo wide local excision breast surgery and SFRT over 60-100 minutes once negative margins are obtained.
  Interventions: Procedure: Therapeutic Conventional Surgery; Radiation: Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Therapeutic Conventional Surgery — Undergo wide local excision breast surgery
Radiation: Radiation Therapy — Undergo SFRT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RT
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well radiation therapy works in treating post-menopausal women with early stage breast cancer undergoing surgery. Radiation therapy uses high energy x rays to kill tumor cells. This may be an effective treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. For select patients with early stage breast cancer undergoing wide local excision followed by single fraction radiation therapy (SFRT), we will evaluate rates of observer-rated toxicity, cosmetic outcomes and patient satisfaction, objective measures of toxicity and quality of life as well as delivery of intended dose.

SECONDARY OBJECTIVE:

I. Locoregional control reported at five years.

OUTLINE:

Patients undergo wide local excision breast surgery and SFRT over 60-100 minutes once negative margins are obtained.

After completion of study treatment, patients are followed at 1 week, 1 month, 3 months, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Core needle biopsy (e.g. Mammotome, core, stereotactic, ultrasound guided) showing invasive mammary cancer (with or without concomitant ductal carcinoma or lobular carcinoma in situ) or ductal carcinoma in situ; acceptable histologic types of invasive mammary cancer include ductal, tubular, mucinous, papillary, cribriform and "NOS" (not otherwise specified); invasive lobular cancer is excluded
* Age >= 50 years and postmenopausal with no menses for at least one year prior to study enrollment
* Age > 70 years with invasive breast cancer clinical size =< 3 cm OR Age 50 - 70 years with invasive breast cancer clinical size =< 1.5 cm OR Age >= 50 years and postmenopausal with any grade ductal carcinoma in situ (DCIS) clinical extent =< 1.5 cm (clinical tumor size will be determined by pre-operative breast imaging-mammography, ultrasound and/or magnetic resonance imaging; in cases of multiple measurements, the largest recorded single dimension will be used to determine eligibility)
* Hormone receptor status

  * Estrogen or progesterone receptor positive or
  * Estrogen and progesterone receptor negative and clinical tumor size =< 1.0 cm
* Human epidermal growth factor receptor 2 (HER2)/neu negative on the core biopsy analysis defined as 0 or 1+ by immunohistochemistry or not amplified by fluorescent in situ hybridization analysis
* Tumor >= 0.5 cm from skin as defined by breast ultrasound
* Unicentric tumor
* Axillary lymph nodes negative by pre-operative physical examination in all cases and pathologic examination from surgery for invasive disease
* Negative surgical margins, defined as no margin-labeling ink on tumor cells from margin evaluation

Exclusion Criteria:

* Initial core biopsy showing invasive lobular cancer
* Estrogen receptor and progesterone receptor negative tumor with clinical size > 1 cm
* Any Her 2+ breast cancer (immunohistochemistry 3+; or amplified by fluorescence in situ hybridization [FISH])
* Cancer in a patient with a known inherited susceptibility mutation in breast cancer (BRCA)1 or BRCA2
* Multicentric breast cancer (two foci of known cancer in the breast separated by greater than 5 cm, or in separate quadrants
* Clinically or pathologically positive axillary lymph nodes
* Any prior breast cancer
* Prior breast radiation therapy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Mattson, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Radiation Therapy)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (Radiation Therapy)
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (NA) — 1 participant
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events as a Measure of Safety and Tolerability
Description: Toxicity will be assessed by the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) v 3.0.
Time Frame: Up to 2 years
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Radiation Therapy)
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Quality-of-life Assessments
Description: Will be rated by patients using the POST-B, the Functional Assessment of Chronic Illness Therapy (FACIT), and the Skindex-16.
Time Frame: Up to 2 years
Population: The study was terminated early by the IRB due to the fact that an IDE (Investigational Device Exemption) was never submitted. No outcome measure data was collected.
Arm/Group | Treatment (Radiation Therapy)
Number analyzed (Participants) | 0

3. Primary Outcome: Cosmetic Differences in the Treated Breast
Description: Will measure differences in the cosmetic size, shape, or texture of the breast. Cosmesis will be graded according to the Baker Scale. Patient reported cosmesis will also be evaluated using the Ontario Clinical Oncology Breast Cancer Questionnaire.
Time Frame: Up to 2 years
Population: as for outcome 2
Arm/Group | Treatment (Radiation Therapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Locoregional Control Rate
Description: Locoregional control will be calculated with confidence interval estimates and will be compared to historical control rates.
Time Frame: At 5 years
Population: as for outcome 2
Arm/Group | Treatment (Radiation Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: The overall survival will be analyzed using Kaplan-Meier method.
Time Frame: Up to 5 years
Population: as for outcome 2
Arm/Group | Treatment (Radiation Therapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: Disease Specific Survival
Description: The disease specific survival will be analyzed using Kaplan-Meier method.
Time Frame: Up to 5 years
Population: as for outcome 2
Arm/Group | Treatment (Radiation Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Radiation Therapy)
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Radiation Therapy) (N=1)
Fibrosis (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast oedema (Reproductive system and breast disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early by the IRB due to the fact that an IDE (Investigational Device Exemption) was never submitted. No outcome measure data was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes